CLINICAL TRIAL: NCT03732521
Title: Clinical, Randomized and Double-blind Controlled Trial of an Educational Therapeutic Intervention for Family Caregivers on the Psychological and Behavioral Symptoms of Dementias (PRESTA Study)
Brief Title: Management of Psychological and Behavioral Symptoms in Patients With Dementias
Acronym: PRESTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CEIC-10/2014
Record Dates: First submitted 2018-10-05; First posted 2018-11-06 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Dementia; Family Relations; Psychological and Behavioral Symptoms
Keywords: Dementia; family caregiver; Zarit scale; NPI-10; psychological and behavioral symptoms
MeSH Terms: conditions — Dementia; Behavioral Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): educational therapy
  Interventions: Other: Educational therapy
- Control group (No Intervention): usual clinical practice

INTERVENTIONS:
Other: Educational therapy — educational intervention to the caregiver and individualization according to their family and social context
  Arms: Intervention group

SUMMARY:
Background: The psychological and behavioral symptoms (SPCD) of dementias are the manifestations that cause the most suffering in the patient and caregiver, worsening the other two symptomatic areas (cognitive and functional) and precipitating the early institutionalization of patients with dementia. non-pharmacological therapies (TNF) in dementia are framed in the biopsychosocial model of patient care. We found evidence in the literature about the effectiveness of ambulatory educational interventions to the family caregiver in terms of reducing overload and improving their state of mind But it is not well demonstrated whether this improvement can have an indirect impact on the SPCD of the patient, nor whether the profile of patients could have an added benefit to the best pharmacological treatment.

Methods: The experimental study selected thirty-six older adults family caregivers of patients with dementia.The intervention group (n=18) received isolated medical treatment, while the control group (n=18) received medical treatment plus educational support therapy to their family caregivers. Data collection included sociodemographic measures and responses to the educational support therapy tot the Zarit Caregiver Overload Scale (family caregivers) and Neuropsychiatric Inventory (NPI-10) patients with dementia.

DETAILED DESCRIPTION:
A descriptive analysis of the sociodemographic characteristics of the intervention and control groups was done. Qualitative variables were expressed as percentages, and quantitative variables were summarised as the median and interquartile range.

Shapiro-Wilk tests indicated that the dependent variables were not normally distributed (p < .05), so non-parametric statistical analyses were subsequently performed. The difference between the medians of the two patient groups was examined with the Mann-Whitney U test. Qualitative variables were compared with the chi-squared or Fisher's exact test, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of at least 6 months of dementia and on treatment with IACEs ± memantine.
* Patients diagnosed with dementia, who score on the global scale of Severity of Reisberg between 4 and 6, both included.
* Patients who at least obtain a score ≥ 4 on the NPI scale, version validated in Spanish. The symptoms must be present at least one month prior to the visit and will not be attributable to intercurrent medical pathology or to acute confusional syndrome.
* Patients living in a family home, and accompanied by a family caregiver who agrees to sign the informed consent after obtaining all the information of the study in question.

Exclusion Criteria:

* Patients with a diagnosis of mild cognitive impairment or who do not take specific medication (IACEs and / or memantine).
* Patients with severe sensory deprivation that does not allow MMSE scale assessment.
* Patients who present intercurrent medical illnesses that confers a poor short-term vital prognosis (6 months).
* Patients in which the SPCD may be in the context of a toxicometabolic disease, uncontrolled pain or delirium, according to the researcher's clinical criteria.
* Patients who are taking typical neuroleptics, long-acting BZD, major opioids or drugs that can potentially alter the state of consciousness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-02-10 (Actual); Primary Completion 2016-11-20 (Actual); Study Completion 2017-09-05 (Actual)

PRIMARY OUTCOMES:
Caregiver Activity Survey (Zarit scale) measures caregiver overload. | At the beginning of the enrolment and 3 months later.
  Change from baseline Zarit scale at 3 months. To assess caregiver burden we use the Zarit scale (Caregiver Overload Scale), validated in our setting and widely used not only in studies of dependency, but also in other populations. It consists of 22 questions with 5 possible answers (never, rarely, sometimes, quite often, quite often, almost always), scored from 1 to 5, and with a range of 22 to 110 in the total score, and which establishes the different degrees of overload according to the score obtained: absence of overload (≤ 46), light overload (47-55) and intense overload (≥ 56). The main drawback to its use is the size and, therefore, the time involved in its use.
Neuropsychiatric Inventory (NPI). | At the beginning of the enrolment and 3 months later.
  Change from baseline of the NPI-10. The Neuropsychiatric Inventory (NPI) 10 items, is a relatively brief interview with a family member or friend who knows the patient well and can evaluate 12 behavioral areas commonly affected in patients with dementia, including depression. It is also routinely used to evaluate the effects of treatment on these symptoms. The total severity score on the NPI-10 represents the sum of the individual symptom scores and ranges from 0 to 36 . Caregiver distress associated with the symptom is scored on a 0- to 5-point anchored scale identical to that used in the NPI.

SECONDARY OUTCOMES:
Sociodemographic measures. | At the beginning of the enrolment.
  Gender (man and woman), Age (years) and Employment status (acoccupationally active or inactive).

CONTACTS AND LOCATIONS:
Locations (1):
- Calamanda Matamoros, Tortosa, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No